CLINICAL TRIAL: NCT03353038
Title: A 3D Printed Assistive Technology Intervention: A Phase I Trial
Brief Title: A 3D Printed Assistive Technology Intervention
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-17-0025
Record Dates: First submitted 2017-11-06; First posted 2017-11-24 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Chronic Disease
Keywords: assistive technology; 3 Dimensional Printing; Self-Management
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Off-The-Shelf Pillbox vs 3D Printed Pillbox (Active Comparator): Participants in the study were pillbox users at baseline. Participants described their experiences and preferences with their own pillbox. Then participants will be given a 3D printed pillbox. Researchers will compare participants' experiences and preferences between their off-the-shelf pillbox used at baseline and the customized 3D printed pillbox delivered to participants as part of the study.
  Interventions: Device: 3D printed pillbox

INTERVENTIONS:
Device: 3D printed pillbox — The research team interviewed the participant about their habits, routines, preferences, medications, and skills and abilities. Based on the interview, the research team designed and printed a customized 3D printed pillbox.

SUMMARY:
The purpose of this study is to understand the feasibility of using a 3D printer to create tailored assistive technology rehabilitation devices. Specifically, we are investigating if a tailored 3D printed pillbox is safe, acceptable, and effective compared to an off-the-shelf generic pillbox. In this study, approximately 20 people with chronic health conditions who use pillboxes will describe their satisfaction and medication adherence with their current pillbox using a series of surveys and interviews. Then they will partake in an interview about their pillbox, medications, and routines. Based on the interview, the research team will 3D print a new pillbox tailored to the participant's preferences, abilities, and medication regimen. Then the participant will use the pillbox for 2-8 weeks. At the end, the participant will answer the same questions describing their satisfaction and medication adherence with the new pillbox using a series of surveys and interviews. This research will reveal important knowledge about the potential of 3D printing in the clinic and effectiveness of customized assistive technology.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Adults (ages 18+ years)
* Use a pillbox at least weekly
* Prescribed 2+ medications
* Willing to try a new 3D printed pillbox

Exclusion Criteria:

* Have significant cognitive impairment evidenced by a score of 10+ on the short blessed test
* Unable to meet with the research team in person and by phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 1 week and again at 2-8 Weeks
  The participant will be asked if they experienced any changes in their health or major issues using their pillbox at 1 week and at the end of the study. Also, all participants were educated to contact to the study team should they experience an adverse event.
Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST2.0) | 2-8 Weeks
  The participant will complete the QUEST 2.0 to describe their satisfaction with the 3D printed pillbox as compared to their satisfaction with the off the shelf pillbox. This will demonstrate the acceptability of the device.
Adherence to Refills and Medications Scale (ARMS) | 2-8 Weeks
  Medication adherence as measured by the ARMS will demonstrate the preliminary efficacy of the of the 3D printed assistive technology. Specifically, it will help determine if the pillbox helped participants better take their medications as prescribed.

IPD SHARING:
Plan to Share IPD: No